CLINICAL TRIAL: NCT06777225
Title: The Effect of Breathing Exercise on Nausea, Vomiting and Anxiety in Patients With Gynecological Cancer Receiving Chemotherapy: Randomized Controlled Study
Brief Title: Breathing Exercise Application in Patients With Gynecological Cancer.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Didem Gül, nurse, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAKU-HEM-DG-01
Record Dates: First submitted 2024-12-31; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Gynecological Cancer
Keywords: nausea; vomiting; gynecological canser; anxiety
MeSH Terms: conditions — Nausea; Vomiting; Anxiety Disorders | interventions — Breathing Exercises; Weights and Measures

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled study. It includes an experimental and a control group.
Who Masked: Participant
Masking Description: It will be checked whether there is a difference between the experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The patient was given detailed information about the research and intervention, and written consent was obtained with an informed consent form.
  The patient's information was obtained through a diagnostic information form containing sociodemographic information.
  1st, 2nd, 3rd Cycle (The following steps were followed.) The Rhodes Nausea Vomiting and Retching Index (BCI), Beck Anxiety Scale and VAS pain scale were applied and evaluated by the researcher.
  The patient was directed to the room determined by the nurse in the outpatient treatment unit.
  Breathing exercises were applied to the patient. The patient's chemotherapy infusion was started. After the patient's chemotherapy was completed, breathing exercises were applied again.
  The post-test was applied. Note: The satisfaction survey was evaluated only after the 3rd cycle.
  Interventions: Other: breathing exercises; Other: scale; Other: scala
- control group (Other): The patient was given detailed information about the research and intervention, and written consent was obtained with an informed consent form.
  The patient's information was obtained through a diagnostic information form containing sociodemographic information.
  1st, 2nd, 3rd Course (The following steps were followed.) The researcher applied the Rhodes Nausea Vomiting and Retching Index (BCOI), Beck Anxiety Scale and VAS pain scale as a pre-test and evaluated the patient.
  The patient was directed to the room determined by the nurse in the outpatient treatment unit.
  The patient's chemotherapy was started. The post-test was applied after the chemotherapy was completed.
  Interventions: Other: scale; Other: scala

INTERVENTIONS:
Other: breathing exercises — This study is to examine the effects of breathing exercises on nausea, vomiting and anxiety levels in patients with gynecological cancer.
  1 Exercise:
  * Find a quiet, calm and comfortable place for yourself.
  * Lie on your back in a comfortable place (flat surface, bed or couch) and bend your knees or sit in a comfortable place (chair or armchair).
  * Close your eyes.
  * Place your left hand on your belly and your right hand on your chest.
  * Take a deep breath through your nose for 4 seconds.
  * Feel your hand on your belly rise and your belly swell as you breathe in.
  * Make sure your chest is not swollen.
  * Hold your breath for 4 seconds. Breathe out in 4 seconds.
  * Do this 10 times every day, morning and evening, 3 times.
  Arms: experimental group
Other: scale — The patient received standard nursing care and the scale was applied after the intervention. The 21-question inventory developed by Dr. Aaron T. Beck was used. The reliability and validity of the Beck Depression Inventory (BDI), which is used to measure the severity of depression, was performed in our country by N. Hisli in 1989. (Cronbach's alpha value was calculated as 0.85). Each question takes a value between 0-3 points. When evaluating the results; 0-10 points are normal; 11-16 points are mild mood disorder; 17-20 points are borderline clinical depression; 21-30 points are moderate depression; 31-40 points are severe depression and over 40 points are very severe depression (Çiçekçe et al, 2023).
  Other Names: Beck anxiety scale
Other: scala — The scale was developed by Rhodes and McDaniel (1999), and its Turkish validity and reliability were carried out by Fatma Genç and Mehtap Tan. The scale, which evaluates the number and severity of nausea-vomiting-retching episodes in the last 24 hours, consists of eight items. The scale has three sub-dimensions: Symptom Experience, Symptom Formation, and Symptom Distress. The responses to the items on the five-point Likert-type scale are scored as 0 = minimum 22 distress level, 4 = maximum distress level. When evaluating the scores, items 1, 3, 6, and 7 are reversed. The highest score that can be obtained from the scale is 32, and higher scores mean that nausea-vomiting symptoms have increased in patients (Odabaşı et al, 2021).
  Other Names: rhodes nausea and vomiting scale

SUMMARY:
The aim of this study is to determine the effects of breathing exercises on nausea, vomiting and anxiety levels in patients with gynecological cancer.

DETAILED DESCRIPTION:
When looking at statistical data, the number of individuals diagnosed with cancer is increasing every year and it is estimated that there will be approximately 30.2 million new cancer cases worldwide in 2040 . When looking at statistical data and literature, it is shown that there is an increase in survival rates thanks to developing technology. Cervix, endometrium, ovary, vulva, vagina and fallopian tube cancers are called gynecological cancers specific to women . According to current data, the incidence rates of gynecological cancers in our country are; endometrium cancer is fifth (5.6%), ovarian cancer is seventh (3.3%) and cervix cancer is ninth (2.3%). Being diagnosed with gynecological cancer is the beginning of a difficult process for every woman. The emotions felt at the time of diagnosis, the process of accepting the cancer diagnosis, and getting oneself together and starting treatment make it difficult to cope. Both the disease and the treatments such as surgery, chemotherapy, and radiotherapy cause patients to experience many serious physical, psychosocial, and sexual symptoms. The symptoms and symptom severity experienced by patients may vary depending on the type, stage, and treatments applied to gynecological cancers. Along with chemotherapy, symptoms such as anxiety, changes in vital signs due to anxiety, depression, weight change, reluctance, apathy, sleep problems, changes in motor and cognitive activities, weakness or loss of energy, inadequate self-care, feeling worthless, guilt, helplessness, hopelessness, thoughts of suicide or death, and inability to concentrate can be observed at varying levels depending on the clinical course of the disease. In summary, the disease process brings with it physical, social, economic and psychological problems and negatively affects the individual's quality of life . Anxiety is a natural reaction that an individual develops against situations in which they do not feel safe. Uncertainty is the most important factor that leads to anxiety. When the uncertainty in the disease experience is evaluated as a danger by the individual, the anxiety experienced increases even more . For this reason, the process experienced by cancer patients due to the disease itself, the toxicity created by the treatment and the symptoms should be evaluated and their anxiety should be defined. In addition to the diagnosis of cancer, symptoms caused by the treatment also increase the anxiety of the cancer patient. When looking at studies conducted with cancer patients, it is reported that patients experience symptoms such as mucositis, pain, nausea and vomiting, anorexia, cachexia, dehydration, taste changes, alopecia, dyspnea, dry mouth, fatigue, immunosuppression and psychological problems . Nausea and vomiting, which are frequently encountered during the treatment process, negatively affect the patient's quality of life and increase their anxiety. Nausea and vomiting resulting from chemotherapy treatment are divided into five groups depending on the time of onset and the type of treatment. Acute nausea and vomiting is defined as nausea and vomiting that occurs within a few minutes or hours following treatment, usually reaches its most severe level in the 5-6th hour and passes within 24 hours, delayed nausea and vomiting occurs after the 24th hour of chemotherapy, mostly within 72 hours and can last for a week in some chemotherapy applications, anticipatory nausea and vomiting occurs during or before chemotherapy, breakthrough vomiting is nausea and vomiting that occurs again within 24 hours after chemotherapy despite the use of the most appropriate prophylactic treatment, and refractory vomiting is defined as nausea and vomiting that the patient has experienced during the previous treatment process, that cannot be prevented as a result of prophylactic antiemetic treatment and that does not respond to additional treatments applied to the patient.

In the study conducted by Farrel et al.; It has been found that the physical functional status, nutritional status and quality of life of patients experiencing nausea and vomiting are negatively affected. It is stated in the literature that in order to control nausea and vomiting, people are increasingly inclined to use non-drug methods such as hypnotherapy, behavioral therapy, breathing exercises, regulation of nutrition and life routines, massage, acupuncture and herbal treatments. In the literature, breathing exercises are among the recommended lifestyle changes to alleviate nausea and vomiting.

It has also been stated that breathing exercises, which are among the independent nursing initiatives of nurses, reduce tension and anxiety caused by stress. Most of the treatments in Western medicine are expressed as general, complementary and alternative medicine. The United States National Health Institute has divided these methods into two basic groups as "natural products" and "body-mind practices". In this context, breathing therapy is a body-mind practice. 'The Regulation on Complementary and Alternative Treatment Practices in our country was published in the Official Gazette on October 27, 2014 with the number 29158 and entered into force'. Today, people attempt to learn breathing techniques due to their positive effects in the treatment of diseases or in the management of their symptoms. Although there is very limited evidence of the healing effects of breath therapy from the past to the present, it is seen that the scientific studies in the literature on women's health and breath therapy have increased in the last decade. The words breath, inhale, exhale are identified with the most basic energy, life energy and creativity needed directly to live in many languages, and this meaning goes beyond the air we breathe. Breath is our primary activity that accompanies us in every area of our lives and enables us to survive in a healthy way for a quality life. When we look at the known history of breath therapy, the healing power of breathing techniques has been the most important treatment method since the beginning of human history. Since it is known that it is possible to affect consciousness and provide physical healing with breathing techniques, in the spiritual and mystical tradition that has continued from ancient times to the present, efforts have been made to create consciousness expansions by triggering the breath with sudden shapes.

When the studies conducted are examined, it has been determined that breathing exercises are effective on anxiety, quality of life, fatigue, pain, nausea, vomiting and vital signs in patients. Studies have shown that anxiety and nausea and vomiting affect each other. It has been observed that when the nausea and vomiting levels of the patients decrease or when their nausea and vomiting pass, their anxiety levels decrease/pass.

Diaphragmatic breathing exercise focuses on slowing down the respiratory rate. The most important aspect of breath control is taking diaphragmatic breaths. Diaphragmatic breathing consists of a smooth and deep breath. It is a breathing technique that uses the contraction of the diaphragm muscle to move the breath downward in the body. Diaphragmatic breathing has been shown to increase vital capacity in patients with asthma and functional capacity in patients with heart failure and chronic obstructive pulmonary disease (COPD). Diaphragmatic breathing exercise, guided imagery and progressive muscle relaxation exercises have been shown to significantly increase physical function and quality of life in patients with breast and prostate cancer. Chest breathing exercise aims to relax by focusing on breathing and breathing slowly and deeply. Chest breathing exercise applied twice a day in gynecological cancer patients receiving chemotherapy has been shown to reduce fatigue. It has been determined that continuous nursing care and chest breathing exercise have a positive effect on respiratory functions, self-care adequacy and sleep duration in patients diagnosed with lung cancer. In studies conducted in our country, breathing exercises are insufficient in patients with gynecological cancer receiving chemotherapy. This study will be conducted to determine nausea, vomiting and anxiety levels by applying breathing exercises to patients with gynecological cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old.

  * Stage 1-2-3.
  * Being literate.
  * Having volunteer patients.
  * Being diagnosed with gynecological cancer.
  * Being a female patient receiving chemotherapy for the first time.
  * Not smoking or consuming alcohol.
  * Will receive 3 cycles of chemotherapy, 21 days apart.
  * Not having a psychiatric diagnosis.

Exclusion Criteria:

* Stage 4.

  * Those who have been diagnosed with cancer but have not received treatment and cannot complete the cure.
  * Those with communication and psychiatric problems.
  * Those who do not know how to read, write and speak Turkish.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients over 18 years old
  1st cycle chemotherapy literate stage1-2-3
Enrollment: 104 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The effect of breathing exercise on nausea, vomiting and anxiety in patients with gynecological cancer receiving chemotherapy: Randomized Controlled Study. | 20 week
  It is planned to be performed in Ankara Etlik City Hospital Adult Outpatient Chemotherapy Unit. The universe will consist of individuals who have been diagnosed with gynecological cancer in the relevant institution, will start their first course of chemotherapy, have stage 1-2-3 cancer, will receive 3 courses of chemotherapy at 21-day intervals, volunteer for the study, are 18 years of age and older, and are literate. In this study, the sample size was calculated with 95% theoretical power using the "G. Power-3.1.9.2" program before data collection. In order to determine whether there was a difference between the experimental and control groups in terms of nausea, vomiting and anxiety due to the breathing exercise applied to gynecological cancer patients receiving chemotherapy, an independent sample t-test was performed based on the two-sided Wilcoxon-Mann-Whitney test for 1:1 group allocation (Faul, 2007). For this reason, Kareem and Afiyanti's studies were taken as reference (Kareem
Effect of breathing exercise on nausea, vomiting and anxiety in gynecological cancer patients receiving chemotherapy: A Randomized Controlled Trial. | 20 week
  Beck Anxiety Inventory
  A 21-question inventory developed by Dr. Aaron T. Beck was used. The reliability and validity of the Beck Depression Inventory (BDI), which is used to measure the severity of depression, was performed in our country by N. Hisli in 1989.
  (Cronbach's alpha value was calculated as 0.85). Each question takes a value between 0-3 points. When evaluating the results; 0-10 points are normal; 11-16 points are mild mood disorder; 17-20 points are borderline clinical depression; 21-30 points are moderate depression; 31-40 points are severe depression and over 40 points are very severe depression (Çiçekçe et al, 2023).
Effect of breathing exercise on nausea, vomiting and anxiety in gynecological cancer patients receiving chemotherapy: A Randomized Controlled Trial. | 20 week
  Rhodes Nausea Vomiting and Retching Scale
  The scale was developed by Rhodes and McDaniel (1999), and its Turkish validity and reliability were made by Fatma Genç and Mehtap Tan. The scale, which evaluates the number and severity of nausea-vomiting-retching in the last 24 hours, consists of eight items. The scale has three sub-dimensions: Symptom Experience, Symptom Formation and Symptom Distress. The responses to the items on the five-point Likert-type scale are scored as 0 = minimum 22 distress level, 4 = maximum distress level. When evaluating the scores, items 1, 3, 6 and 7 are reversed.
  The highest score that can be obtained from the scale is 32, and higher scores mean that nausea-vomiting symptoms have increased in patients (Odabaşı et al, 2021).

CONTACTS AND LOCATIONS:
Overall Officials: Didem Gül,graduate student, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Etlik şehir hastanesi, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No